CLINICAL TRIAL: NCT06031961
Title: A Double-blind Randomized Placebo - Controlled Trial of Oral Melatonin as Premedication Agent in Pediatrics Undergoing Therapeutic Cardiac Catheterization
Brief Title: The Premedication Properties of Oral Melatonin in Pediatrics Undergoing Therapeutic Cardiac Catheterization
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hussein Ali, lecturer in anesthesiology department, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Melatonin in PA
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Anesthesia
Keywords: Melatonin, premedication, preoperative anxiety
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1st group: Melatonin group (Active Comparator): All children in this group have to receive 0.5 mg/kg of melatonin(maximum dose 20 mg) which will be administered orally on the night before surgery ( at 12 am) and immediately before 30 minutes before entering the catheterization room.
  Interventions: Drug: melatonin
- 2nd group: Placebo group (Placebo Comparator): All children in this group have to receive a placebo which will be administered orally on the night before surgery and immediately before 30 minutes before entering the catheterization room.
  Interventions: Drug: melatonin

INTERVENTIONS:
Drug: melatonin — We will premedicate the children whom involved in the 1st group with 0.5 mg/kg oral melatonin in the midnight before surgery and the dose will be repeated at morning before getting in the catheterization room
  Other Names: Placebo

SUMMARY:
The evaluation of oral melatonin efficacy as premedicant agent in pediatrics undergoing elective cardiac interventions is the primary outcomes of our trail.

DETAILED DESCRIPTION:
About 65 % of children whom undergoing surgery and anesthesia are suffering from keen anxiety and stress especially in the preoperative holding area. This situation mostly extends to the parents and this can worse the child response before surgery. The intensity of child anxiety had been reported to be a powerful predictor for incidence of hallucination in the recovery period and new-onset unpleasant behavioral changes such as nightmares and enuresis. In general, patients' preoperative anxiety if not controlled or reduced by premeditations, it can influence the surgical outcomes such as the postoperative pain, analgesic requirements, length of hospitality. Many of systemic physiological changes may be associated with the anxiety; such as elevated respiratory rate, elevated blood pressure, increased the heart rate and developing the risky of arrhythmia; all of these can be dilemmas and obstacles in the way of the anesthesiologist in choosing the appropriate method of anesthesia or the appropriate drugs for the starting and continuation of anesthesia. At the beginning of the eighties of the last century, the midazolam had been presented as the finest oral premedication agent which used in the pre-operative period for children to reduce the anxiety, and its quickly achieved wide acceptance as the preferred primer before induction of anesthesia. Rapid absorption during oral administration, multiple route administration and low incidence of nausea with its use when compared with other benzodiazepines, all these features helped to favor the midazolam for pre-operative use as a premedication in pediatrics. Despite the decent advantages that midazolam has in use before surgical interventions as a premedication agent, especially for children, it has some drawbacks that may affect the results of the surgical procedure and the anesthesia plan. Paradoxical reactions, interaction with opioids, overdue evacuation during the recovery time and capricious bioavailability are the most common drawbacks of midazolam in general. Some of these effects of midazolam had been shown to vary with patient age. In the presence of such drawbacks with the use of midazolam, the emergence of a suitable alternative may be widely accepted. Naturally, the N-acetyl-5-methoxy-tryptamine, which is also known as the Melatonin, is a biogenic amine which is firstly discovered in the middle of last century (1958) by Aaron B. Lerner in Yale University. After a while, the melatonin had been reported to be synthesized in animals, plants and even in unicellular organisms such as bacteria. In humans, the melatonin is mainly produced by the bovine pineal glands which is a small pine-cone shaped structure and located on the roof of the 3rd ventricle, deeply within the brain. In addition to production of melatonin; the main function of pineal gland; the gland also secrets some substances such as Oxytocin, Serotonin and Orexin in responding to influencing by neurotransmitters from neurons and nerve cells. The lymphocytes, bone marrow, eyes, and the gastrointestinal tract had been recently documented to a site production of melatonin hormone in human body.

Sleep cycle, mood, memory dreaming, immune activity, learning fertility and reproduction are the common physiological activities which regulated mainly by the melatonin in humans, all of these functions are accomplished through direct stimulation or binding to melatonin receptors.

European Medicines Agency had licensed the synthetic melatonin in form of tablets (2 mg) and (3 mg) in United Kingdom (UK) and Hungary. Also there is a licensed oral solution of 1mg/ml. The unlicensed synthetic melatonin is available in different forms from Kidmel® & Kidnaps®, Special Products Limited in the UK in liquid formulations and capsule formulation of 2 & 3 mg.

Many qualities of the chemical melatonin, which is mostly produced by the pineal gland, may help explain why it has cardio protective benefits. Melatonin may have receptor-mediated or receptor-independent protective effects. Ischemia/reperfusion (IR) injury has been shown to affect many organs, including the heart, liver, kidney, gut, testis, brain, and lung. Melatonin has been shown to offer numerous protective advantages. Melatonin's potent antioxidant qualities, as well as its capacity to encourage the synthesis of other antioxidants such as glutathione reductase, catalase, glutathione peroxidase, and superoxide dismutase, all contribute to its protective effects.

As a result, it acts as both an indirect antioxidant and a free radical scavenger. Because melatonin receptors are found in the vasculature, it is possible that melatonin has local control over cardiovascular diseases. Furthermore, the amount of melatonin generated by persons suffering from coronary artery disease is inversely connected to the stage of the disease-the less melatonin produced, the more advanced the disease.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4-12 years.
* scheduled for elective therapeutic cardiac catheterization
* ASA I and II

Exclusion Criteria:

* ASA III or more than.
* Drug allergy.
* Any of contraindication for general anesthesia.
* Mental and neurological diseases.
* disapproval or dissatisfaction
* Liver disease
* Diabetic children
* Thyroid storm
* Sleep disorders
* Intake of antipsychotics.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-09-10 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
preoperative anxiety | 30 minutes before 2nd dose of premedication, 1 hour after 2nd dose premedication, At separation from parents, 5 minutes before induction of general anesthesia.
  Modified Yale Preoperative Anxiety Scale (mYPAS)

SECONDARY OUTCOMES:
Sedation level | 1 hour after 2nd dose premedication, At separation from parents, 5 minutes before induction of general anesthesia.
  The University of Michigan Sedation Scale (UMSS)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed kahloul, professor, Study Chair — souse university
Locations (1):
- Ministry of Health, Baghdad, Thi-Qar, Iraq

IPD SHARING:
Plan to Share IPD: No